CLINICAL TRIAL: NCT04384185
Title: Effectiveness of a Therapeutic Exercise Protocol Combined With Manual Therapy Techniques on the Diaphragm Muscle in Patients With Low Back Pain
Brief Title: Combined Treatment of Manual Therapy and Therapeutic Exercise in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, PhD. Daniel Pecos Martín, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/12
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain, Mechanical; Musculoskeletal Manipulations; Exercise Training
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Exercise therapy (Experimental): Group A: will perform an exercise protocol to improve the stability of the spine muscle of low-back
  Interventions: Other: Exercise protocol
- Group B. Manual therapy and exercises (Experimental): Group B: Will be treated with manual therapy in the diaphragm muscle and the same protocol of therapeutic exercise applied in group A
  Interventions: Other: Exercise protocol; Other: Manual therapy

INTERVENTIONS:
Other: Exercise protocol — Exercises:
  * Pelvic tilt.
  * brinding.
  * cuadruped arm/leg raise.
  * Abdominal strengthening exercises.
  * Low-back muscles stretching.
  * The side bridge.
  * Side leg separation
Other: Manual therapy — 1. Functional diaphragm balancing technique: gentle vertical pressure was applied for 5 minutes at the diaphragm level.
  2. Muscle fiber stretching technique: a cranial traction was performed from the lower edge of the costal arches during the inspiratory breathing phase, for more than 10 respiratory cycles.
  3. Phrenic-center inhibition technique (Figure 3C): the soft tissue was pumped during the expiratory phase by gently and simultaneously using both hands to create pressure in cranial and caudal direction, for more than 10 respiratory cycles.
  Other Names: Myofascial manipulation
  Arms: Group B. Manual therapy and exercises

SUMMARY:
MAIN OBJECTIVE: to assess whether an exercise protocol on the lumbar musculature by adding manual therapy techniques on the diaphragm muscle has the same or greater effect on chronic non-specific lumbar pain than an isolated exercise protocol.

SECONDARY OBJECTIVES: to evaluate the effectiveness of a lumbar exercise protocol in chronic non-specific low back pain in isolation; To evaluate the effectiveness of both therapies in improving joint range in patients with chronic non-specific low back pain and, finally, to assess catastrophism and the avoidance of lumbar mobility when carrying out loaded movements.

HYPOTHESIS: that a lumbar exercise protocol combined with manual therapy treatment on the diaphragm is equal or more effective on pain in patients with chronic nonspecific low back pain than treatment with the same lumbar exercise protocol in isolation.

DETAILED DESCRIPTION:
METHODOLOGY: A prospective randomized clinical trial with two types of intervention (lumbar exercise protocol and manual diaphragm therapy) will be carried out. The variables to be measured are pain, disability, mobility and kinesiophobia. It will be performed in two groups of 21 people who are of legal age, who have low back pain of more than 3 months duration and which is of non-specific origin.

The patients will be randomized and divided into two groups A (control) and B (experimental).

Group A will undergo an exercise protocol.

Group B will undergo the same protocol plus manual therapy techniques on diaphragm muscle. Study participants will have treatment twice a week for 8 weeks, the first information session and the second measurement-evaluation session in the first week of treatment. In the following 3 weeks the session will last 40 minutes for both groups. In the 4th week the established measurements will be carried out again.

ELIGIBILITY:
Inclusion Criteria:

* Legal age
* Non-specific Low-Back pain
* Pain more 3 months

Exclusion Criteria:

* subjects with lumbar herniation.
* Spine canal stenosis
* Subjects with neurological disease.
* Lumbar surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Low-back pain | Change from Baseline disability at 3 months
  The investigators use a Visual Analog Scale (VAS) to determine the intensity of the patient with lowback pain.The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and ten the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.

SECONDARY OUTCOMES:
Disability with Oswestry Disability Index | Change from Baseline disability at 3 months
  The Oswestry Disability Index (ODI) is a questionnaire used by clinicians and researchers to quantify disability for low back pain.The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible
Lumbar range of motion | Change from Baseline disability at 3 months
  Mobility. It will be measured using an electronic inclinometer.The TiltMeter© -advanced level and inclinometer app is an inclinometer app of iPhone®. The investigation has demonstrated that the app possesses good to excellent reliability (ICC ≥ 0.77) and concurrent validity with a gravity-based inclinometer (r ≥ 0.86) for measuring standing isolated lumbar flexion and extension range of movement
Kinesiophobia | Change from Baseline disability at 3 months
  Kinesiophobia was measured by an 11-item version of the Tampa Scale of Kinesiophobia (TSK-11). The 11 items of the scale each have 4 response options; all anchored with the answers "strongly disagree", which scores 1 point, and "strongly agree", which scores 4 points. The total sum score is calculated and can range between 11 and 44 points. A high score indicates strong fear of movement/(re)injury, i.e. high kinesiophobia. TSK-11 has been psychometrically evaluated and has shown good construct validity and reliability among older people (i.e. internal consistency (Cronbach alpha, 0.74-0.87) and test-retest reliability (ICC r = 0.747)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego Izquierdo, PhD, Study Chair — Alcala University
Locations (1):
- Grupo Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain